CLINICAL TRIAL: NCT05867719
Title: The Physiological Effects of Acute and Ramp Simulated Altitude Exposure During Simulated Flight Tasks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Texas, El Paso (Other)
Responsible Party: Principal Investigator, Jeffrey Eggleston, Assistant Professor of Kinesiology, University of Texas, El Paso
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2042946-1
Record Dates: First submitted 2023-04-13; First posted 2023-05-22 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Altitude Hypoxia
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normoxic (No Intervention): Participants will complete three flight simulator tasks at a normoxic (baseline) altitude. During the flight simulator, participants will need to accomplish three tasks: 1) Maintaining an altitude of 5,000 ft of elevation while performing a mental math test, 2) Flying the aircraft through the center of a series of 7 targets, and 3) Taking off and flying the aircraft a short distance to land on the center of an indicated target.
- Simulated 8,000 feet hypoxic (Experimental): Participants will complete three flight simulator tasks at a simulated 8,000 foot altitude. During the flight simulator, participants will need to accomplish three tasks: 1) Maintaining an altitude of 5,000 ft of elevation while performing a mental math test, 2) Flying the aircraft through the center of a series of 7 targets, and 3) Taking off and flying the aircraft a short distance to land on the center of an indicated target.
  Interventions: Other: Hypoxic breathing conditions
- Simulated 12,000 feet hypoxic (Experimental): Participants will complete three flight simulator tasks at a simulated 12,000 foot altitude. During the flight simulator, participants will need to accomplish three tasks: 1) Maintaining an altitude of 5,000 ft of elevation while performing a mental math test, 2) Flying the aircraft through the center of a series of 7 targets, and 3) Taking off and flying the aircraft a short distance to land on the center of an indicated target.
  Interventions: Other: Hypoxic breathing conditions
- Ramp hypoxic exposure (Experimental): Participants will complete three flight simulator tasks in a ramp exposure breathing at simulated 8,000 feet for five minutes before ascending to simulated 12,000 feet while flying in a flight simulator. During the flight simulator, participants will need to accomplish three tasks: 1) Maintaining an altitude of 5,000 ft of elevation while performing a mental math test, 2) Flying the aircraft through the center of a series of 7 targets, and 3) Taking off and flying the aircraft a short distance to land on the center of an indicated target.
  Interventions: Other: Hypoxic breathing conditions

INTERVENTIONS:
Other: Hypoxic breathing conditions — Participants will undergo three separate hypoxic conditions, along with a normoxic condition, simulating 8,000 foot elevation, 12,0000 foot elevation, and a ramp condition starting at 8,000 feet and then ascending to 12,000 feet.
  Arms: Ramp hypoxic exposure; Simulated 12,000 feet hypoxic; Simulated 8,000 feet hypoxic

SUMMARY:
• The purpose of this study is to investigate which physiological process that controls normal human body homeostasis is affected by low levels of acute hypoxic exposure and whether there is a difference in those physiological processes and simulated flight performance between a rapid and ramp hypoxic exposure. To accomplish this, pilot analogs will be exposed to normoxic, simulated 8,000 ft (2438 m), simulated 12,000 ft (3658 m), and a ramp exposure breathing at simulated 8,000 ft for 5 minutes before ascending to simulated 12,000 ft while flying in a flight simulator. During the flight simulator, participants will need to accomplish three tasks: 1) Maintaining an altitude of 5,000 ft of elevation while performing a mental math test, 2) Flying the aircraft through the center of a series of 7 targets, and 3) Taking off and flying the aircraft a short distance to land on the center of an indicated target. Physiological measures of heart rate variability (HRV), blood pressure (BP), peripheral oxygen saturation (SpO2), electrodermal activity (EDA), and neck neuromuscular activity using electromyography (EMG) will be measured for this study. Along with questionnaires to assess hypoxic symptoms, simulator sickness, and self-perceived workload for each task

ELIGIBILITY:
Inclusion Criteria:

* Meets body composition standards for the US Navy Active-duty personnel based on height and weight
* Normal vision/corrected to normal vision

Exclusion Criteria:

* Respiratory Deficiencies
* Cardiovascular Disorders
* Neurological/Musculoskeletal Disorders
* Photosensitive Epilepsy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Flight performance | 10 minutes per each of the 4 conditions
  ability to perform in-flight assigned tasks
Self-perceived workload | 1 minute to complete the survey, 3 times per condition for 4 conditions
  NASA TLX survey
Electrodermal activity | 10 minutes per each of the 4 conditions
  electrical characteristics of the skin observed as changes in the resistance of the skin to a small electrical current

IPD SHARING:
Plan to Share IPD: No